CLINICAL TRIAL: NCT00898378
Title: Cancer Care Engineering of Colorectal Cancer - OMICs Pilot Study
Brief Title: Study of Biomarkers in Blood & Tissue Samples From Patients With Colorectal Cancer or Polyps & Patients Without Polyps
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0808-24; IUCRO-0221; P30CA082709 (NIH); IUCRO-0221 (Other: Indiana University Cancer Center)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Colorectal Cancer; Healthy, no Evidence of Disease; Precancerous Condition
Keywords: healthy, no evidence of disease; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent rectal cancer; recurrent colon cancer; adenomatous polyp
MeSH Terms: conditions — Colorectal Neoplasms; Precancerous Conditions; Colonic Neoplasms; Rectal Neoplasms; Adenomatous Polyps | interventions — Gene Expression Profiling; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis; Chromatography, Gas; Chromatography, Liquid; Mass Spectrometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens will be analyzed to study metabolimics, lipidomics, genomics, glycoproteomics, global proteomics and Vitamin D status.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Colorectal Cancer Patients: Patients with stages I/II, III and IV colorectal cancer
  Interventions: Genetic: gene expression analysis; Genetic: polymerase chain reaction; Genetic: polymorphism analysis; Genetic: protein expression analysis; Genetic: proteomic profiling; Other: gas chromatography; Other: laboratory biomarker analysis; Other: liquid chromatography; Other: mass spectrometry; Other: questionnaire administration
- Colorectal Polyps Patients: Patients with adenomatous polyp(s) after colonoscopy.
  Interventions: Genetic: gene expression analysis; Genetic: polymerase chain reaction; Genetic: polymorphism analysis; Genetic: protein expression analysis; Genetic: proteomic profiling; Other: gas chromatography; Other: laboratory biomarker analysis; Other: liquid chromatography; Other: mass spectrometry; Other: questionnaire administration
- Healthy Controls: No abnormalities after colonoscopy.
  Interventions: Genetic: gene expression analysis; Genetic: polymerase chain reaction; Genetic: polymorphism analysis; Genetic: protein expression analysis; Genetic: proteomic profiling; Other: gas chromatography; Other: laboratory biomarker analysis; Other: liquid chromatography; Other: mass spectrometry; Other: questionnaire administration

INTERVENTIONS:
Genetic: gene expression analysis — gene expression analysis
Genetic: polymerase chain reaction — polymerase chain reaction
Genetic: polymorphism analysis — polymorphism analysis
Genetic: protein expression analysis — protein expression analysis
Genetic: proteomic profiling — proteomic profiling
Other: gas chromatography — gas chromatography
Other: laboratory biomarker analysis — laboratory biomarker analysis
Other: liquid chromatography — liquid chromatography
Other: mass spectrometry — mass spectrometry
Other: questionnaire administration — questionnaire administration

SUMMARY:
RATIONALE: Studying samples of blood and tissue in the laboratory from patients with cancer, patients with colorectal polyps and from patients without polyps may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at biomarkers in blood and tissue samples from patients with colorectal cancer or colorectal polyps and from patients without polyps (healthy volunteers).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Perform metabolomic, lipidomic, glycoproteomic, proteomic, and genomic (OMIC) profiling using blood and tissue samples from patients with colorectal cancer (CRC) or colorectal adenomatous polyps and from patients without polyps.
* Create an OMIC profile to predict the risk of CRC based on differences observed between patients with CRC, patients with colorectal adenomatous polyps, and patients without polyps.

Secondary

* Create an OMIC profile to predict response and toxicity to specific chemotherapies, biological therapies, and radiotherapy for CRC.
* Utilize a novel knowledge discovery tool (BioMap) based on literature mining and, in the future, utilize the results of the OMIC analyses to identify interactive molecular pathways that underlie the development and progression of CRC.

OUTLINE: Patients with locally advanced or metastatic colorectal cancer are stratified according to treatment (first-line chemotherapy with fluorouracil [5-FU]/oxaliplatin or 5-FU/irinotecan vs second- or third-line chemotherapy with irinotecan only vs biological therapy with bevacizumab vs biological therapy with cetuximab vs radiotherapy).

Blood and tissue samples are collected periodically for laboratory studies. Samples are analyzed for metabolomics by nuclear magnetic resonance, gas chromatography, liquid chromatography, and mass spectrometry; lipidomics, proteomics, and glycoproteomics by liquid chromatography and mass spectrometry; and genomics (single nucleotide polymorphism biomarkers) by PCR. Vitamin D status is also assessed.

Patients complete diet-history and lifestyle questionnaires at baseline and once a year for 2 years. Healthy volunteers complete these questionnaires only at baseline.

After completion of study, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter. Healthy volunteers are not followed after study completion.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Diagnosis of one of the following:

    * Stage I or II colorectal cancer (CRC)*

      * Planning to undergo surgery only
    * Stage III CRC*

      * Planning to undergo surgery followed by adjuvant chemotherapy with or without neoadjuvant chemoradiotherapy
    * Stage IV CRC

      * Planning to undergo chemotherapy and biologic therapy (bevacizumab, cetuximab, or panitumumab)
    * Colorectal adenomatous polyps

      * Planning to undergo colonoscopy
  * Healthy volunteer

    * Planning to undergo colonoscopy NOTE: *Patients with previously resected stage II or III CRC are eligible provided they undergo blood sample collection prior to starting chemotherapy

PATIENT CHARACTERISTICS:

* Not pregnant
* Able to undergo an 8-hour overnight fast prior to metabolomic testing
* Able to attend follow-up or treatment visits for up to 24 months for collection of blood samples
* No prior or concurrent invasive cancer other than CRC (for patients with CRC)
* No prior invasive cancer and no first-degree relative with a known history of CRC (for healthy volunteers and patients with colorectal polyps)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited via oncology, gastroenterology and surgical oncology clinics at Indiana University Medical Center. Healthy controls will be subjects without any abnormalities after a colonoscopy. Subjects with polyps will be those whose colonoscopy identifies adenomatous polyps (informed consent will be signed first and samples will be collected; after colonoscopy the samples will be identified as "healthy" or "polyps").
Sampling Method: Non-Probability Sample
Enrollment: 551 (Actual)
Dates: Start 2009-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Metabolomic, lipidomic, glycoproteomic, proteomic, and genomic (OMIC) profiling | End of Study
Creation of an OMIC profile to predict the risk of colorectal cancer (CRC) | End of Study

SECONDARY OUTCOMES:
Creation of an OMIC profile to predict response and toxicity to specific therapies for CRC | End of Study
Identification of interactive molecular pathways that underlie the development and progression of CRC | End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Loehrer, MD, Principal Investigator — Indiana University Melvin and Bren Simon Cancer Center
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States